CLINICAL TRIAL: NCT00586859
Title: Multi-Center Study of the NDO Surgical Plicator Utilizing Multiple Implants
Brief Title: Multi-Center Study of the NDO Surgical Plicator Utilizing Multiple Implants for the Treatment of GERD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsoring company ceased business operations.
Sponsor: NDO Surgical, Inc. (Industry)
Responsible Party: Bruce Gaumond, Associate Director, Clinical Affairs, NDO Surgical
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 135-02420
Record Dates: First submitted 2007-12-21; First posted 2008-01-07 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: GERD
Keywords: Gastroesophageal Reflux Disease (GERD); NDO Full-thickness Plicator; Plicator; Endoluminal GERD Therapy
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): NDO Full-thickness Plicator Procedure
  Interventions: Device: NDO Full-thickness Plicator

INTERVENTIONS:
Device: NDO Full-thickness Plicator — The Plicator and gastroscope assembly were passed into the stomach. The stomach was distended with air. The gastroscope was advanced and retroflexed so that the instrument could be visualized and accurately positioned. The Plicator was retroflexed to within 1cm below the GE junction, and the helical tissue retractor was advanced deeply into the gastric wall. The gastric wall was retracted into the Plicator instrument arms. The arms were then closed, and the suture-implant was deployed to secure the full-thickness plication. The tissue retractor is then disengaged and the suture-implant released from the instrument. Additional sutures were placed in the same manner described above, with each additional implant placed incrementally closer to the GE junction in a linear configuration along the anterior gastric cardia. All plications were placed de novo, and re-treatment was not permitted.

SUMMARY:
The purpose of this study was to evaluate the safety and efficacy of placing multiple transmural sutures for the treatment of GERD.

A prospective, multi-center, open-label trial was conducted at four centers in Germany to evaluate a modified Plicator technique for the treatment of patients with symptomatic GERD. Primary efficacy was based on analysis of the GERD Health Related Qualify of Life (HRQL) questionnaire at 6-months post-treatment. Additional efficacy outcomes assessed were heartburn and regurgitation symptoms scores, visual analog scale (VAS) score, GERD medication use, esophageal pH/manometry, and esophagitis. Trial sample size was chosen to provide 87% power in detecting a 50% median reduction in GERD-HRQL score at an alpha level of 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* History of heartburn or regurgitation for at least 6 months.
* Esophageal manometry study (conducted within the previous 6 months) demonstrating an adequate resting pressure of the lower esophageal sphincter (LES) of at least 5 mm Hg.
* pH study (conducted within the previous 6 months) demonstrating pathological reflux (defined as the total % time of pH<4.0 > 4.5% or a DeMeester composite score > 14.7).
* Symptoms requiring daily PPI therapy.
* GERD-HRQL scores must be > 15 while Off Medication and Off Medication scores must be > 6 points higher than On-Medication scores.
* Subject is a surgical candidate in the event of a complication related to this procedure, Class ASA I or II.
* Subject agrees to participate and signs consent form.

Exclusion Criteria:

* Patient is pregnant.
* Patient has hiatal hernia > 3 cm.
* Presence of persistent dysphagia, weight loss, esophageal bleeding, vomiting (>1 per week) or gas/bloat.
* Esophagitis grades III or IV by Savary criteria.or type C or D by Los Angeles classification .
* Barrett's esophagus with dysplasia.
* Patient has had a previous endoscopic (Endocinch, Stretta, Enteryx, etc.) or surgical repair (Nissen Fundoplication, etc.) performed to treat GERD.
* Active medical condition that would preclude the subject from finishing this study.
* Abnormal blood coagulation or the chronic use of anticoagulant or platelet anti-aggregation therapy (other than for cardiac prophylaxis).
* Pathological changes in soft tissue that would prevent secure fixation of the EPS Implant.
* Presence of esophageal or gastric varices.
* Esophageal dysmotility as determined by manometry studies.
* Esophageal stricture.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2006-05; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
GERD Health Related Qualify of Life (HRQL) questionnaire at 6-months post-treatment | 1, 6, 12, 24, 36, 48 and 60-month post-treatment

SECONDARY OUTCOMES:
Heartburn Score | 1, 6, 12, 24, 36, 48 and 60-months post-treatment
Regurgitation score | 1, 6, 12, 24, 36, 48 and 60-months post-treatment
GERD symptom improvement as measured by a visual analog scale | 1, 6, 12. 24, 36, 48 and 60-months post-treatment
GERD medication use | 1, 6, 12, 24, 36, 48 and 60-months post-treatment
Esophageal acid exposure | 6-months post-treatment
Esophageal sphincter (LES) resting pressure as measure by manometry | 6-months post-treatment
Esophagitis score | 6-months post-treatment

CONTACTS AND LOCATIONS:
Locations (4):
- Germany (4):
  - Evangelisches Krankenhaus, Düsseldorf
  - Markus-Krankenhaus, Frankfurt
  - Medizinische Klinik und Poliklinik Universitatsklinikum Leipzig, Leipzig
  - Klinikum Ludwigsburg, Ludwigsburg